CLINICAL TRIAL: NCT00957866
Title: Prospective Anti-HCV Trial of Peg-Interferon and Ribavirin in Subjects of First Nations, Metis and Caucasian Ethnicity: PRAIRIE Study
Brief Title: Prospective Anti-Hepatitis C Virus (Anti-HCV) Trial of Peg-Interferon and Ribavirin in Subjects of First Nations, Metis and Caucasian Ethnicity
Acronym: Praire
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Minuk G, Head of department, Section of Hepatology, Health Sciences Centre, John Bhuler Centre.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B2008:164
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Hepatitis C
Keywords: The number of cases in the database thus far (4,477) is clearly sufficient to achieve meaningful results
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Pegylated Interferons (Peg-IFN) and Ribavirin — A anti-viral regimen with a combination of pegylated Interferons (Peg-IFN) and Ribavirin

SUMMARY:
Background:

According to recent estimates, the prevalence of Chronic Hepatitis C (CHC) in Canada is three times more common in First Nations (FN)and Metis compared to non-FN populations. Moreover, once infected, the progression of CHC to cirrhosis and/or hepatocellular carcinoma is greater in FN patients due to the increased prevalence of alcohol abuse, obesity and diabetes in this segment of the population.

Research Plan:

This research proposal consists of three parts. The objective of Part I is to document the response to anti-viral treatment for CHC among treatment-naïve FN and Metis and Caucasian (hereafter referred to as non-FN) patients residing in three urban Western Canadian centres (Winnipeg, Saskatoon and Regina). Demographic, clinical and response to treatment data in a total of 160 patients (80/group) will be collected at the above centres and transferred to the Section of Hepatology at the University of Manitoba for statistical analyses. In Part II, the applicants will document and compare the immune responses to HCV proteins throughout the course of therapy in FN, Metis and non-FN patients. In the final part, direct economic costs of CHC care in FN, Metis and non-FN patients will be ascertained and future costs predicted.

Hypotheses:

Part I - The rate of sustained virologic response (SVR) to treatment for CHC is higher in FN and Metis compared to non-FN and no Metis patients.

Part II - The immune response to HCV proteins during anti-viral therapy for CHC is enhanced in FN and Metis compared to non-FN and non-Metis patients.

Part III - The direct costs of health care utilization and delivery for CHC are similar among FN and Metis and non-FN and non- Metis patients.

DETAILED DESCRIPTION:
Specific Objectives:

1. To provide detailed information on the demographics and clinical characteristics of treatment-naïve FN and Metis versus non-FN and Non-Metis patients proceeding to treatment for CHC.
2. To document and compare SVR and sustained biochemical response (SBR) rates, adherence to therapy, side effects, dose adjustments and discontinuation of treatment between FN and Metis and non-FN and Non-Metis patients.
3. To determine whether the immunologic features associated with SVR (increased NK cell activity and enhanced interferon gamma production by CD4 cells in response to viral antigens) differ in FN and Metis and non-FN and non-Metis patients.
4. To document and compare the direct costs of health care utilization and delivery for CHC between FN and Metis and non-FN and Non-Metis patients.
5. Develop a model predicting outcome of therapy, using demographic, clinical and viral characteristics, and test the model with race as one of the explanatory variables.
6. To forecast future prevalence, mortality and medical costs of CHC care in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of FN and metis and non-FN descent referred for treatment at the three centres will be candidates for this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
SVR is the primary outcome for this study. SVR is defined as a negative serum HCV-RNA by a qualitative test sensitive to <50 IU/ml six months after the completion of therapy14, performed by a Health Canada approved laboratory. | 3years

CONTACTS AND LOCATIONS:
Overall Officials: Minuk Gerald, MD, Principal Investigator — University of Manitoba, Health Science senter
Locations (3):
- Canada (3):
  - The University of Manitoba, Winnipeg, Manitoba
  - University of Regina, Regina, Saskatchewan
  - University of Saskatchewan, Saskatoon, Saskatchewan